CLINICAL TRIAL: NCT04525573
Title: Effects of a Red/Gold/IR LED Combination Light on Reduction of Fat
Status: Withdrawn | Type: Observational
Why Stopped: Lost principal investigator. Have not picked up a new PI yet.
Sponsor: Ward Photonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CP20-01
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Body Image; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Testing:
  * Glucose
  * CMP
  * A1c
  * Fructosamine
  * Lipids
  * Leptin
  * CRP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: LLLT Combination Red/Gold/IR Therapy — Three LLLT combination treatments per week over the course of two consecutive weeks, and a final follow up on day-15 (total of 7 treatments).

SUMMARY:
An open-label evaluation of the effects of a red/gold/IR LED combination light on reduction of fat. The results shall be compared to previous results from a comparator device utilizing only red LED monotherapy for the non-invasive reduction in fat layer for body contouring.

DETAILED DESCRIPTION:
The combination of gold/red/IR light is theorized to enhance the effect of the deeper penetrating red/IR light with the photomodulated effects of gold light. The light is positioned alongside the patient as they lay, or sit on a treatment table. A light panel is mounted to an articulating arm for positioning the light at the correct treatment position above the patient (non-contact). The effects of a red/gold/IR combination LED light therapy device on circumferential reduction of fat will be measured, and the overall health of the patients will be monitored using blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is 18 years of age or older.
* Diagnosed with adult-onset (type 2) diabetes.
* Obesity

Exclusion Criteria:

* Photosensitive condition or medication.
* Active chemotherapy treatment or other cancer treatment.
* Pregnant, possibly pregnant or planning pregnancy prior to the end of study participation.
* Developmental disability or cognitive impairment that, in the opinion of the investigator, would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Chronic stomach conditions (IBS, Crohn's, Ulcerative Colitis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women over the age of 18 and with diagnosed Type 2 diabetes who are seeking fat loss.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fat Reduction | 15 days
  Circumferential reduction of fat as measured around the observation areas of the body.

SECONDARY OUTCOMES:
General Health Improvement | 15 days
  The secondary outcome of this study is to monitor patient health changes during the treatment period. The principal method for monitoring patient health is through blood testing. There is some evidence in literature that patients undergoing fat reduction benefit from secondary effects associated with their general health.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsaraf Dabawala, MD, Principal Investigator — Horizon Medical Center
Locations (1):
- Horizon Medical Center, Schaumburg, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study is an open-label evaluation of the effects of a red/gold/IR LED combination light on reduction of fat. And general health of the patients will be monitored as a possible correlation with fat reduction. However, the findings from this study are intended to explore whether a larger comparative study should be conducted.

REFERENCES:
- [Background] Opel DR, Hagstrom E, Pace AK, Sisto K, Hirano-Ali SA, Desai S, Swan J. Light-emitting Diodes: A Brief Review and Clinical Experience. J Clin Aesthet Dermatol. 2015 Jun;8(6):36-44. PMID 26155326
- [Background] Lee SY, Park KH, Choi JW, Kwon JK, Lee DR, Shin MS, Lee JS, You CE, Park MY. A prospective, randomized, placebo-controlled, double-blinded, and split-face clinical study on LED phototherapy for skin rejuvenation: clinical, profilometric, histologic, ultrastructural, and biochemical evaluations and comparison of three different treatment settings. J Photochem Photobiol B. 2007 Jul 27;88(1):51-67. doi: 10.1016/j.jphotobiol.2007.04.008. Epub 2007 May 1. PMID 17566756
- [Background] Goldberg DJ, Amin S, Russell BA, Phelps R, Kellett N, Reilly LA. Combined 633-nm and 830-nm led treatment of photoaging skin. J Drugs Dermatol. 2006 Sep;5(8):748-53. PMID 16989189
- [Background] Sadick NS. A study to determine the efficacy of a novel handheld light-emitting diode device in the treatment of photoaged skin. J Cosmet Dermatol. 2008 Dec;7(4):263-7. doi: 10.1111/j.1473-2165.2008.00404.x. PMID 19146602
- [Background] Baez F, Reilly LR. The use of light-emitting diode therapy in the treatment of photoaged skin. J Cosmet Dermatol. 2007 Sep;6(3):189-94. doi: 10.1111/j.1473-2165.2007.00329.x. PMID 17760698
- [Background] Russell BA, Kellett N, Reilly LR. A study to determine the efficacy of combination LED light therapy (633 nm and 830 nm) in facial skin rejuvenation. J Cosmet Laser Ther. 2005 Dec;7(3-4):196-200. doi: 10.1080/14764170500370059. PMID 16414908
- [Background] Lee SY, You CE, Park MY. Blue and red light combination LED phototherapy for acne vulgaris in patients with skin phototype IV. Lasers Surg Med. 2007 Feb;39(2):180-8. doi: 10.1002/lsm.20412. PMID 17111415
- [Background] Goldberg DJ, Russell BA. Combination blue (415 nm) and red (633 nm) LED phototherapy in the treatment of mild to severe acne vulgaris. J Cosmet Laser Ther. 2006 Jun;8(2):71-5. doi: 10.1080/14764170600735912. PMID 16766484
- [Background] Sadick N. A study to determine the effect of combination blue (415 nm) and near-infrared (830 nm) light-emitting diode (LED) therapy for moderate acne vulgaris. J Cosmet Laser Ther. 2009 Jun;11(2):125-8. doi: 10.1080/14764170902777349. PMID 19391058
- [Background] Kwon HH, Lee JB, Yoon JY, Park SY, Ryu HH, Park BM, Kim YJ, Suh DH. The clinical and histological effect of home-use, combination blue-red LED phototherapy for mild-to-moderate acne vulgaris in Korean patients: a double-blind, randomized controlled trial. Br J Dermatol. 2013 May;168(5):1088-94. doi: 10.1111/bjd.12186. PMID 23278295
- [Background] Ablon G. Combination 830-nm and 633-nm light-emitting diode phototherapy shows promise in the treatment of recalcitrant psoriasis: preliminary findings. Photomed Laser Surg. 2010 Feb;28(1):141-6. doi: 10.1089/pho.2009.2484. PMID 19764893